CLINICAL TRIAL: NCT01361672
Title: Attain Ability® Family Left Ventricular Lead Chronic Performance Study
Brief Title: Model 4296 Left Ventricular (LV) Lead Chronic Performance Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 4296 Chronic Performance
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lead survivability will be summarized.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate long-term performance of the 4296 LV Lead. This evaluation is based on the number of lead-related complications occurring during the study compared to the number of leads enrolled in the study. The leads will be followed for 5 years after implant. This study is required by FDA as a condition of approval of the Model 4296 LV Lead. This study is conducted within Medtronic's post-market surveillance platform.

ELIGIBILITY:
Patients who meet all of the following inclusion criteria and do not meet any of the following exclusion criteria are eligible for enrollment.

Inclusion Criteria

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive an Attain Ability Model 4296 LV lead
* Patient within 30 day post implant enrollment window

Exclusion Criteria

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a 4296 LV Lead within 30 days. All subjects must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Model 4296 LV Lead-related complication rate | 5 years
  To demonstrate that the Model 4296 lead-related complication-free probability

SECONDARY OUTCOMES:
Types of lead-related adverse device effects | 5 years
  To summarize all lead related adverse events
Percent of subjects with changes in electrode programming | 5 years
  To characterize any changes in electrical programming
Number of fractures with and without loss of function | 5 years
  To characterize fractures with and without loss of function
Bipolar electrical performance at 1 year | 1 year
  To summarize bipolar electrical performance at one year post implant
Bipolar pacing impedance | 1 year
  To characterize threshold measurements and impedance for both conductors
Bipolar pacing capture threshold | 1 year
  To characterize standard bipolar pacing voltage thresholds

CONTACTS AND LOCATIONS:
Locations (99):
- United States (94):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Chandler, Arizona
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Monterey, California
  - Rancho Mirage, California
  - Redding, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Safety Harbor, Florida
  - Tampa, Florida
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Hyattsville, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Marquette, Michigan
  - Ypsilanti, Michigan
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Morristown, New Jersey
  - Ocean City, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - Huntington, New York
  - New York, New York
  - Poughkeepsie, New York
  - Utica, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Allentown, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Falls Church, Virginia
  - Leesburg, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (4):
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Essen, Germany